CLINICAL TRIAL: NCT05123716
Title: Drug Effects on Interpersonal Interaction
Acronym: DEI
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: IRB21-0778
Record Dates: First submitted 2021-11-05; First posted 2021-11-17 (Actual); Last update posted 2022-06-15 (Actual); Status verified 2022-06

CONDITIONS: Interaction, Social
MeSH Terms: interventions — N-Methyl-3,4-methylenedioxyamphetamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Experimental: Placebo Then MDMA (Experimental): Participants first receive placebo at their first session in the laboratory. Then will return to the laboratory 72 hours later and will receive 100 mg MDMA.
  Interventions: Drug: MDMA; Drug: placebo oral tablet
- Experimental: MDMA Then Placebo (Experimental): Participants first receive 100 mg MDMA at their first session in the laboratory. Then will return to the laboratory 72 hours later and will receive placebo.
  Interventions: Drug: MDMA; Drug: placebo oral tablet

INTERVENTIONS:
Drug: MDMA — Participants will be given 100 mg of MDMA
Drug: placebo oral tablet — Participants will be given a placebo capsule that will only contain lactose.

SUMMARY:
The investigators propose to use a Paired Partner design, in which subjects engage in a 45-min semi-structured conversation with one (novel) partner under the influence of MDMA and with another partner under the influence of placebo. At the end of each session, they will rate their feelings about the partner, and on the test day, subjects will be asked which partner they preferred and felt closer to.

DETAILED DESCRIPTION:
The study will use a within-subject design with three sessions: i) MDMA and conversation with Person A, ii) placebo and conversation with Person B, iii) test session (online) assessing preference for Persons A and B. The MDMA dose will be 100 mg, administered under double blind conditions. The conversation will consist of a 45 min dialog between the participant and the partner, a person trained to engage in conversation for this purpose. The dyad will be provided with topics to discuss, at their own pace. The order of administration of drug and placebo will be counterbalanced, and the partners will be same-sex and varied across sessions. The primary outcome measures will be feelings of closeness and connection at the end of the two drug sessions, at the online test session and follow-up. After study completion, participants will be fully informed about the study.

ELIGIBILITY:
Inclusion Criteria:

* English fluency
* High school level education
* BMI between 19 and 30

Exclusion Criteria:

* Diagnosed medical condition
* women who are nursing, pregnant, or plan to become pregnant within 3 months
* History of psychotic disorder or family history of psychotic disorder

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2022-05-01 (Actual); Study Completion 2022-05-01 (Actual)

PRIMARY OUTCOMES:
Profile of Mood States | Time Frame: Baseline-72 hours after completion of the sessions
  The POMS measures individuals' mood states. This is a validated scale to measure positive and negative mood states. The POMS contains 30 items and assesses six identified mood factors: Tension-Anxiety, Depression-Ejection, Anger- Hostility, Vigor-Activity, Fatigue-Inertia, and Confusion-Bewilderment. Scoring of the instrument provides a global score of 0 to 120 or individual domain scores. Lower scores indicate better mood state. The POMS brief form is a simple self-rating instrument.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Undecided